CLINICAL TRIAL: NCT05830552
Title: The Effect of Feedback on Physical Activity Surveillance Using Wearable Device-Smartphone Application for Resolution of Metabolic Syndrome in Aged 60 or Older ; a 12-Week Randomized Control Study
Brief Title: The Effect of Feedback on Physical Activity Surveillance Using Wearable Device-Smartphone Application for Resolution of Metabolic Syndrome in Aged 60 or Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Young Jin Tak, Principal Investigator, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PNUHH-2109-021-107
Record Dates: First submitted 2023-03-21; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Metabolic Syndrome; Physical Activity; Wearable Device
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: In the intervention group, the researcher provided feedback on the participants' exercise amount through telephone contact every two weeks during the 12-week study period. It includes recommendations for continuing exercise therapy based on the recommendations for physical activity. Through phone consultations, they answered questions about exercise or discussed problems, were encouraged to continue exercising, answered questions or discussed problems related to wearable devices and apps, and encouraged for continuous data transmission.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the intervention group, the researcher gave feedback on the subjects' exercise amount through telephone contact every 2 weeks during the 12-week study period. Through phone consultations, they answered questions about exercise or discussed problems, encouraged to continue exercising, answered questions or discussed problems related to wearable devices and encouraged continuous data transmission.
  Interventions: Other: Receving feedback
- Control Group (Placebo Comparator): In the case of the control group, physical activity is monitored by itself through wearable devices and smartphone apps without phone counseling.
  Interventions: Other: No regular feedback

INTERVENTIONS:
Other: Receving feedback — Receving regular feedback from a health provider
  Arms: Intervention Group
Other: No regular feedback — No regular feedback from a health provider
  Arms: Control Group

SUMMARY:
The Effect of Feedback on Physical Activity Surveillance using Wearable Device-Smartphone Application for Resolution of Metabolic Syndrome in Aged 60 or older; a 12-Week Randomized Control Study

DETAILED DESCRIPTION:
Research on whether wearable device interventions can effectively prevent metabolic syndrome remains insufficient. This study aimed to evaluate the effect of feedback on clinical indicators in patients with metabolic syndrome aged 60 or older on activities measured using wearable devices, such as smartphone apps. Patients aged 60 or older diagnosed with metabolic syndrome were recruited and prescribed to survive for 12 weeks using wrist-worn devices (B.BAND, B Life Inc, Korea). The block randomization method was used to distribute the participants between an intervention group (n=20) and control group (n=20). In the intervention group, an experienced study coordinator provided feedback on physical activity to individuals through telephone counseling every other week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with metabolic syndrome by a doctor.
* Aged 60 or older.
* A person who understands the clinical trial process and signs the consent form
* Possession of a smartphone and a daily mobile phone user for the past 3. months and expected to use for more than 3 months.
* A person who agrees to provide the data on the amount of physical activity measured and collected by a wearable device.
* A person who can exercise at an intensity more than walking for 12 weeks.

Exclusion Criteria:

* Under the aged 60.
* A person who does not agree to provide data on physical activity.
* Those who who are judged to have difficulty in exercising such as walking due to uncontrolled diabetes, high blood pressure or serious cardiovascular disease.
* A person who is not used to or is reluctant to use a smartphone app.
* Those who have difficulty wearing wearable devices due to skin diseases around their wrists.
* A person who is expected to have an unintended change in weight over the next three months due to current pregnancy and planning, thyroid disease, cancer, etc.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in fasting blood tests at baseline and 12th week visits | Baseline and 12th week
  Blood samples were collected from the Jeonju vein after fasting for 6 hours and analyzed in our hospital's laboratory. The lipid profile was tested using an automated analyzer (Hitachi 747, Hitachi Corp, Japan) and enzyme colorimetric method.
Changes in blood pressure (systolic blood pressure, diastolic blood pressure) at baseline and 12th week visits | Baseline and 12th week
  Blood pressure was measured in a sitting position after resting using BP-203 RVII(Colin Corp, Aichi, Japan).
Changes in waist circumference (cm) at baseline and 12th week visits | Baseline and 12th week
  The waist circumference was evaluated by a trained examiner (after normal exhalation) to the nearest millimeter from the midpoint between the lower edge of the rib and the iliac ridge.
Measurement of physical activity through wearable devices | For 12 weeks
  Investigators provided with wrist-wearable device (B.BAND, B Life Inc, Korea), which allowed them to wear and live for 12 weeks. Researchers who have been granted access can check and track participants' physical activity on a daily basis through a web page.

SECONDARY OUTCOMES:
Changes in body weight at baseline and 12th week visits | Baseline and 12th week
  Body weight in kilograms were measured using a digital scale and stadiometer (BSM370, Biospace Co Ltd, Seoul).
Changes in height at baseline and 12th week visits | Baseline and 12th week
  Height in meters were measured using a digital scale and stadiometer (BSM370, Biospace Co Ltd, Seoul).
Changes in body composition at baseline and 12th week visits | Baseline and 12th week
  Body composition was measured by bioelectrical impedance analysis (Inbody 720, Biospace Co Ltd, Seoul)
Depression index at baseline and 12th week visits | Baseline and 12th week
  All participants completed the Beck Depression Inventory (BDI) questionnaires.
Stress scale questionnaires at baseline and 12th week visits | Baseline and 12th week
  All participants completed the Perceived Stress Scale (PSS) questionnaires.
Pulse wave velocity measurement on baseline and 12th week visits | Baseline and 12th week
  Pulse wave velocity was measured in a comfortable supine position using the VP-1000 plus (Omron Healthcare, Bannockburn, IL).

OTHER OUTCOMES:
Gathering subject information from the survey | Baseline
  All participants received information on demographics, occupation (usually for estimating physical activity intensity), frequency and duration of physical activity, history (diagnosis or drug treatment of hypertension, diabetes or dyslipidemia), health-related habits (smoking, drinking and alcohol), and medications taken through the survey. Participants were defined as non-smokers, past smokers, and current smokers, and non-smokers (0 to 98 g/week) or drinkers who drink an average of 7 cups of men and 5 or more cups of women twice per person.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hospital, Busan, Seo-gu, South Korea